CLINICAL TRIAL: NCT05006664
Title: A Phase II Open Label Study of Brentuximab Vedotin in Combination With CHEP in Patients With Previously Untreated CD30-expressing Peripheral T-cell Lymphomas (PTCL)
Brief Title: Brentuximab Vedotin in Combination With CHEP in Patient With PTCL
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Czech Lymphoma Study Group (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CLSG-PTCL-CHEPA
Record Dates: First submitted 2021-08-09; First posted 2021-08-16 (Actual); Last update posted 2021-09-01 (Actual); Status verified 2021-08

CONDITIONS: Lymphoma, T-Cell, Peripheral
Keywords: CD30-expressing; brentuximab vedotin; CHEP
MeSH Terms: conditions — Lymphoma, T-Cell, Peripheral | interventions — Brentuximab Vedotin; Injections; Cyclophosphamide; Doxorubicin; Etoposide; Prednisone

STUDY DESIGN:
Intervention Model Description: Open label, single arm, combination - brentuximab vedotin+cyclophosphamide+doxorubicin+etoposide+prednison
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Brentuximab Vedotin (Adcetris) in Combination with CHEP (Experimental): Single arm, open label, Brentuximab Vedotin (Adcetris) in Combination with CHEP
  Interventions: Drug: Adcetris 50 MG Injection; Drug: Endoxan; Drug: Doxorubicin; Drug: Etoposide; Drug: Prednisone tablet

INTERVENTIONS:
Drug: Adcetris 50 MG Injection — Treatment by study drug Brentuximab Vedotin (Adcetris) in combination with CHEP.
  Other Names: Brentuximab Vedotin
Drug: Endoxan — Treatment by study drug Cyclophosphamide (Endoxan) in combination.
  Other Names: Cyclophosphamide
Drug: Doxorubicin — Treatment by study drug Doxorubicin in combination.
  Other Names: Doxorubicin Ebewe; Doxorubicin Medac
Drug: Etoposide — Treatment by study drug Etoposide in combination.
  Other Names: Etoposide ACCORD
Drug: Prednisone tablet — Treatment by study drug Prednisone in combination.
  Other Names: Prednison Léčiva

SUMMARY:
A Phase II Open Label Study of Brentuximab Vedotin in Combination with CHEP in Patients with Previously Untreated CD30-expressing Peripheral T-cell Lymphomas (PTCL)

DETAILED DESCRIPTION:
Efficacy assessments will be made according to the revised response criteria for malignant lymphoma based on the guidelines of the Lugano Classification (as reported by Cheson B et al. 2014) and will be based on investigator assessment Efficacy will be evaluated in terms of CR rate, ORR, PFS, EFS, OS.

The safety and tolerability of study treatment will be evaluated by means of AE reports (nature, severity, frequency, causality), performance status, physical examinations, ECG and laboratory safety evaluations.

ELIGIBILITY:
Inclusion Criteria:

1. Age >18 years
2. Written informed consent
3. Histologically confirmed diagnosis of CD30-expressing PTCL. The following histological subtypes according to the Revised European-American Lymphoma World Health Organization (WHO) 2016 classification are eligible:

   1. Systemic anaplastic large cell lymphoma (ALCL) ALK+ with age-adjusted international prognostic index (aaIPI) ≥1
   2. Systemic anaplastic large cell lymphoma (ALCL) ALK-
   3. Peripheral T-cell lymphoma not otherwise specified (PTCL-NOS)
   4. Angioimmunoblastic T-cell lymphoma (AITL)
   5. Adult T-cell leukaemia/lymphoma (ATLL; acute and lymphoma types only, must be positive for human T cell leukaemia virus 1)
   6. Enteropathy-associated T-cell lymphoma (EATL)
   7. Hepatosplenic T-cell lymphoma
   8. Monomorphic epitheliotropic intestinal T-cell lymphoma (MEITCL)
   9. Indolent T-cell lymphoproliferative disorder (T-LPD) of the gastrointestinal (GI) tract
   10. Follicular T-cell lymphoma
   11. Nodal peripheral T-cell lymphoma with T-follicular helper (TFH) phenotype
4. Positive CD30 expression by local pathology assessment.
5. Patients must have at least one measurable disease site. The lesion must be fluorodeoxyglucose (FDG)-avid by PET and must have a greatest transverse diameter of ≥1.5 cm and greatest perpendicular diameter of ≥1.0 cm by CT, as assessed by the site radiologist.
6. Eastern Cooperative Oncology Group (ECOG, Appendix B) performance status of 0 to 1
7. Patient must be autologous stem cell transplant (ASCT)-eligible
8. Patient must be appropriate candidate for treatment with anthracyclines
9. Patient must have the following laboratory criteria at screening:

   1. Absolute neutrophil count (ANC) ≥ 1.0 x 109/L (unless secondary to bone marrow involvement by PTCL)
   2. Platelet count ≥ 50 x 109/L (unless secondary to bone marrow involvement by PTCL)
   3. Total serum bilirubin < 1.5 × upper limit of normal (ULN) unless secondary to Gilbert's syndrome or documented liver involvement by lymphoma. Patients with Gilbert's syndrome or documented liver involvement by lymphoma may be included if their total bilirubin is ≤3 × ULN
   4. Alanine transaminase (ALT), aspartate aminotransferase (AST) and alkaline phosphatase (ALP) ≤3 × ULN, or <5 × ULN in cases of documented liver involvement by lymphoma
   5. Serum creatinine clearance must be >40 mL/minute/1.73m2 either measured or calculated using a standard Cockcroft and Gault formula (Cockroft and Gault, 1976, Appendix A) and serum creatinine must be <175 µmol/L.
10. Females of childbearing potential (FCBP) must not be pregnant or breastfeeding and must agree to use at least two effective contraception method during the study and for 6 months following the last dose of treatment.
11. Male participants must: Males who have partners of childbearing potential must agree to use an effective contraceptive method during the study and for 6 months following the last dose of treatment.
12. In the opinion of investigator, the patient must:

    1. be able to understand, give written informed consent, and comply with all study-related procedures, medication use, and evaluations
    2. not have a history of noncompliance in relation to medical regimens or be considered potentially unreliable and/or uncooperative

Exclusion Criteria:

1. Current diagnosis of any following lymphomas:

   1. Primary cutaneous CD30-positive T-cell lymphoproliferative disorders and lymphomas. Cutaneous ALCL with extracutaneous tumour spread beyond locoregional lymph nodes is eligible (previous single-agent treatment to address cutaneous and locoregional disease is permissible)
   2. Mycosis fungoides (MF), including transformed MF
   3. PTCL CD30-negative
2. History of another primary invasive cancer, hematologic malignancy, or myelodysplastic syndrome that has not been in remission for at least 3 years. Exceptions are malignancies with a negligible risk of metastasis or death (e.g., 5-year OS ≥90%), such as carcinoma in situ of the cervix, non- melanoma skin carcinoma, localized prostate cancer, ductal carcinoma in situ, or Stage I uterine cancer.
3. History of progressive multifocal leukoencephalopathy (PML).
4. Known central nervous system (CNS) lymphoma involvement
5. Prior treatment with brentuximab vedotin.
6. Baseline peripheral neuropathy ≥Grade 2 (per the NCI CTCAE, Version 5.0)
7. Left ventricular ejection fraction (LVEF) of < 45% or history of myocardial infarction ≤6 months, or symptomatic cardiac disease (including symptomatic ventricular dysfunction, symptomatic coronary artery disease, and symptomatic arrhythmias) or prior treatment with anthracyclines.
8. Any uncontrolled Grade 3 or higher (per the National Cancer Institute's Common Terminology Criteria for Adverse Events, NCI CTCAE Version 5.0) viral, bacterial, or fungal infection within 2 weeks prior to the first dose of study treatment.
9. Known human immunodeficiency virus (HIV) infection, hepatitis B surface antigen-positive status, or known or suspected active hepatitis C infection.
10. History of hypersensitivity to any component of CHEP, to compounds of similar biological or chemical composition as brentuximab vedotin, and/or the excipients contained in any of the drug formulations of study treatment.
11. Females who are pregnant or breastfeeding
12. Planned CNS prophylaxis with intravenous high-dose methotrexate.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Estimated)
Dates: Start 2021-10 (Estimated); Primary Completion 2024-10 (Estimated); Study Completion 2024-10 (Estimated)

PRIMARY OUTCOMES:
PET-negative complete response (CR) rate at the end of treatment | 6m months
  Complete response

SECONDARY OUTCOMES:
Type, incidence, severity, seriousness, and relatedness of treatment emergent adverse events. | 38 months
  Type, incidence, severity, seriousness, and relatedness of treatment emergent adverse events.
Type, incidence, severity, seriousness, and relatedness of adverse events in the follow-up period. | 38 months
  ype, incidence, severity, seriousness, and relatedness of adverse events in the follow-up period.
Progression-free survival (PFS) | 12 months, 24 months
  PFS is defined as the time from C1D1 to the date of the first clinically or radiologically or histologically/cytologically documented disease progression or death due to any cause. If a patient has not progressed, relapsed, or died as of the clinical cut-off date for final analysis, PFS will be censored on the date of last disease assessment when the patient is known to be alive and progression-free. If no tumour assessments are performed after the baseline visit or all post-baseline tumour assessment results have overall responses of "not evaluable", PFS will be censored on the date of study entry.
  Kaplan Meier plots will be used to estimate the distribution of PFS. The PFS probabilities at 12 and 24 months, and the associate 95% CI will be summarized.
Overall survival (OS) | 12months, 24 months,
  Overall survival (OS) is defined as the time from C1D1 until death from any cause and documented by the date of death.
  Kaplan Meier plots will be used to estimate the distribution of OS. The OS probabilities at 12 and 24 months, and the associate 95% CI will be summarized for each treatment arm.
Event-free survival (EFS) | 12months, 24 months,
  EFS is defined as the time from C1D1 to the date of the first clinically or radiologically documented disease progression or death due to any cause or start of new anti-lymphoma treatment (pre-planned radiotherapy or pre-planned HDT with ASCT are not counted as an event). If a patient has not progressed, relapsed, or died or started a new anti-lymphoma treatment at the analysis cut-off date, EFS will be censored on the date of last contact.
  Kaplan Meier plots will be used to estimate the distribution of EFS. The EFS probabilities at 12 and 24 months, and the associate 95% CI will be summarized.
Objective Response Rate (ORR) at the end of treatment | 38 months
  The ORR is defined as the proportion of patients with CR or PR based on the response achieved at the end of treatment.
  The ORR along with 95% CI will be presented. The number and percentage of patients with CR and the number of patients with PR will also be presented.
Rate of pre-planned upfront HDT/ASCT | 38 months
  The rate of pre-planned upfront HDT/ASCT is defined as the proportion of patients who underwent the pre-planned HDT/ASCT after end of treatment.
  The rate of pre-planned upfront HDT/ASCT along with 95% CI will be presented.
Duration of response (DoR) | 38 months
  Duration of response (DoR) is defined as the time from the date of the first occurrence of a documented CR or PR to the date of disease progression, relapse or death from any cause (PFS), as assessed by the investigator for the subgroup of patients with the CR or PR assessment at EoT evaluation. For patients achieving a response who have not experienced disease progression, relapse, or died prior to the time of the analysis, the duration of response will be censored on the date of last disease assessment.
  Kaplan Meier plots will be used to estimate the distribution of DoR.

CONTACTS AND LOCATIONS:
Overall Officials: Magdaléna Zikmundová, MD, Ph.D., Study Director — Subinvestigator, Protocol completation
Locations (7):
- Czechia (7):
  - University Hospital Brno, Brno
  - University Hospital Hradec Králové, Hradec Králové
  - University Hospital Olomouc, Olomouc
  - University Hospital Ostrava, Ostrava
  - University Hospital Plzeň, Pilsen
  - University Hospital Kralovske Vinohrady, Prague
  - Charles University General Hospital, Prague

IPD SHARING:
Plan to Share IPD: No